CLINICAL TRIAL: NCT02016287
Title: Sequential Paclitaxel Chemotherapy and Radiotherapy as First Line Treatment for Elderly Metastatic Esophageal Squamous Cell Cancer:: a Phase II Single Center Prospective Clinical Trial
Brief Title: Sequential Paclitaxel Chemotherapy and Radiotherapy as 1st Line Treatment for Elderly Esophageal Squamous Cell Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shen Lin (Other)
Responsible Party: Sponsor-Investigator, Shen Lin, Professor, Peking University
Organization: Peking University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGOG7002; CGOG7002 (Registry Identifier: CGOG)
Record Dates: First submitted 2013-12-07; First posted 2013-12-19 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-12

CONDITIONS: Esophageal Squamous Cell Cancer; Elderly Patients
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- sequential treatment (Experimental): paclitaxel treatment and radiotherapy
  Interventions: Other: Sequential chemotherapy （paclitaxel 80mg/m2 d1,d8) and radiotherapy

INTERVENTIONS:
Other: Sequential chemotherapy （paclitaxel 80mg/m2 d1,d8) and radiotherapy — Sequential paclitaxel chemotherapy and radiotherapy

SUMMARY:
Elderly patients with metastatic esophageal squamous cell carcinomas have poor prognosis and majority of them were intolerable to combined chemotherapy in China. In the investigators phase II clinical trial proceeded before, the paclitaxel treatment showed good tolerance and efficacy to esophageal squamous cell carcinomas. Radiotherapy has been indicated as a definitive treatment for unresectable or medically inoperable tumors in ESCC patients. However, not only the combination with chemotherapy, but also the boundaries of the clinical target volume (CTV) are not internationally defined. The investigators then initiated a prospective phase II clinical trial with sequential paclitaxel/cisplatin and radiotherapy as the 1st line treatment in elderly metastatic esophageal carcinoma to observe the efficacy and safety of the combination.

ELIGIBILITY:
Inclusion Criteria:

1. Having signed informed consent Age more than 69 years old
2. Histologically confirmed esophageal squamous carcinoma,metastatic disease with primary tumor,no prior palliative chemotherapy;
3. No prior radiotherapy except radiotherapy at non-target lesion of the study more than 3 months
4. Sex is not limited
5. Measurable disease according to the RECIST criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 15 days before enrollment)
6. Karnofsky performance status ≥80
7. Life expectancy of ≥ 3 month
8. WBC > 3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet > 100,000/mm3, Hb > 9g/dl(within 14 days before enrollment),ALT and AST < 1.5 times ULN (≤5 times ULN in patients with liver metastases),Bilirubin level < 1.0 times ULN,Serum AKP < 2.5 times ULN,Serum creatinine < 1.0 times ULN
9. No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever > 38℃；
10. Normal ECG and heart function
11. Fertile patients must use effective contraception Good compliance

Exclusion Criteria:

1. Previous treatment of palliative chemotherapy
2. Known hypersensitivity to Paclitaxel,Cisplatin
3. Only with Brain or bone metastasis
4. No measurable lesions, eg. pleural fluid and ascites
5. Suffer from severe heart disease or disease with other important organs Chronic diarrhea or renal dysfunction
6. Other previous malignancy within 5 year, except non-melanoma skin cancer
7. Mentally abnormal or disable cognition,including CNS metastasis

Min Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 1 year
  the follow-up visit of PFS will be performed every 2 cycles

SECONDARY OUTCOMES:
overall survival | 2 years
  OS means that from the first dose of treatment drug to death or lost, the follow-up visit will be performed every 3 months till death or lost

OTHER OUTCOMES:
disease control rate | 1 year
adverse events | 2 years
quality of life | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking Universtiy Cancer Hospital
Locations (1):
- Peking University Cancer Hospital, Beijing, Beijing Municipality, China